CLINICAL TRIAL: NCT04165603
Title: Fluorescence-navigated Thoracoscopy for Detection of Small Pulmonary Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018PHB144-01
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5mg/kg of ICG, 24h before surgery (Active Comparator): 5mg/kg of indocyanine green, intravenously injection 24 hours before surgery
  Interventions: Procedure: Preoperative Infusion of Indocyanine Green
- 1mg/kg of ICG, 24h before surgery (Experimental): 1mg/kg of indocyanine green, intravenously injection 24 hours before surgery
  Interventions: Procedure: Preoperative Infusion of Indocyanine Green
- 5mg/kg of ICG, 48h before surgery (Experimental): 5mg/kg of indocyanine green, intravenously injection 48 hours before surgery
  Interventions: Procedure: Preoperative Infusion of Indocyanine Green
- 1mg/kg of ICG, 48h before surgery (Experimental): 1mg/kg of indocyanine green, intravenously injection 48 hours before surgery
  Interventions: Procedure: Preoperative Infusion of Indocyanine Green

INTERVENTIONS:
Procedure: Preoperative Infusion of Indocyanine Green — preoperatively infuse indocyanine green through peripheral vein

SUMMARY:
Fluorescence-navigated thoracoscopic imaging with indocyanine green (ICG) is a novel technique for detection of small pulmonary nodules other than traditional radiography or intraoperative palpation. As a non-targeted fluorescent contrast agent, ICG accumulates in tumors by the enhanced permeability and retention effect (EPR), making the lesions fluoresce under fluorescent imaging. However, the optimal dosage and injection time of ICG are still under exploration. Hence, we perform this study in humans made up of four groups to determine the optimal time and dose.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral pulmonary solid nodules, with diameter 1-3 cm.
* Suitable for surgery and signed informed consent.

Exclusion Criteria:

* Liver dysfunction.
* Allergic to indocyanine green.
* Can't tolerate thoracoscopic surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Signal-to-background Ratio (SBR) of the Tumor and Normal Parenchyma | within 1 week after surgery
  We use image analysis software ImageJ to evaluate the strength of luminosity in tumors and normal parenchyma using intraoperative images and calculate signal-to-background-ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jun, MD, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China